CLINICAL TRIAL: NCT05511597
Title: Turning Around Freezing: Effect of Split-belt Treadmill Training on Daily-life Turning-related Freezing of Gait in Parkinson's Disease
Brief Title: Split-belt Treadmill Training for Freezing of Gait in Parkinson's Disease
Acronym: SBT FOG-TRAIN
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Alice Nieuwboer, Full Professor, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: S65984
Record Dates: First submitted 2022-08-18; First posted 2022-08-23 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Parkinson Disease; Freezing of Gait; Split-belt Treadmill
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Randomised single-blind parallel-group study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants receive training in both arms and will be blinded to the exercise group differences.
  Outcomes assessor will be blinded to the group allocation and will carry out all assessments in a standardized manner irrespective Investigator will perform blinded analyses of the data
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SBT+CP (Experimental): Split-belt training + complex task practice
  Interventions: Behavioral: Split-belt treadmill training; Behavioral: Complex task practice
- SBT+PL (Active Comparator): Split-belt training + static exercise
  Interventions: Behavioral: Split-belt treadmill training; Behavioral: Static balance exercise

INTERVENTIONS:
Behavioral: Split-belt treadmill training — Split-belt walking with various speed ratios between the two legs, applied with random-block practice
Behavioral: Complex task practice — Overground gait flexibility training with added cognitive tasks
  Arms: SBT+CP
Behavioral: Static balance exercise — Mindfulness and breathing combined with static balance exercises
  Arms: SBT+PL

SUMMARY:
A split-belt treadmill (SBT) is a treadmill with two belts, whereby each leg can be driven at a different speed. Previous work by the investigators showed that one session of SBT training improved turning while multi-tasking and reduced FOG in PwPD tested in the laboratory. However, subsequent work raises questions as to whether treadmill improvements following repeated SBT training generalize to overground situations in the long term. Therefore, in this study, the investigators will perform a four-week SBT intervention with added practice of everyday turning scenarios (SBT+CP) or placebo exercise (SBT+PL), and study its effects on FOG in both the laboratory and at home.

ELIGIBILITY:
* Be between 40 - 90 years of age
* Have a diagnosis of Parkinson's disease
* Be able to walk for 10 min without an aid
* Be able to follow and understand the oral instructions of the investigator
* Have a disease stage of I to IV (while ON-medication)
* Have had no change in your Parkinson's medication in the past month (or to your deep brain stimulator if applicable) and also no planned changes in medication over the next 4 months
* Have at least about 1 "freezing" episode per day (based on the New Freezing of Gait Questionnaire: N-FOG)
* Not participating in another clinical trial
* Have no acute joint disease
* Not have any other condition that affects your walking pattern or prevents you from completing all study tasks
* Have not undergone major surgery or hospitalization in the last 3 months
* No substance abuse
* No depressive disorder or other apathetic disorder that precludes daily exercise

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-12-16 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage Time Frozen during turning in place | up to 8 weeks post intervention
  Percentage Time Frozen scored from video of rapid alternating full turns in place. Based on earlier work showing immediate effects of SBT training on FOG during this task.
Time to complete Timed Up and Go (TUG) | up to 8 weeks post intervention
  Overall time to complete the Timed Up and Go task. The training is expected to improve multiple transitions between straight walking and turning and should be reflected in the overall task time.

SECONDARY OUTCOMES:
Percentage Time Frozen over all FOG-provoking tasks | up to 8 weeks post intervention
  Percentage Time Frozen scored from videos of Turning in place,TUG, Hotspot door and Hotspot personalized.
Percentage Time Frozen over 1-week free-living monitoring | up to 8 weeks post intervention
  Percentage Time Frozen estimated from machine learning algorithm using free-living sensor data captured over 1 week.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Nieuwboer, PhD, Principal Investigator — KU Leuven
Locations (1):
- Faculty of Movement and Rehabilitation Sciences (FaBeR), Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] D'Cruz N, Seuthe J, De Somer C, Hulzinga F, Ginis P, Schlenstedt C, Nieuwboer A. Dual Task Turning in Place: A Reliable, Valid, and Responsive Outcome Measure of Freezing of Gait. Mov Disord. 2022 Feb;37(2):269-278. doi: 10.1002/mds.28887. Epub 2021 Dec 22. PMID 34939224
- [Background] D'Cruz N, Seuthe J, Ginis P, Hulzinga F, Schlenstedt C, Nieuwboer A. Short-Term Effects of Single-Session Split-Belt Treadmill Training on Dual-Task Performance in Parkinson's Disease and Healthy Elderly. Front Neurol. 2020 Sep 30;11:560084. doi: 10.3389/fneur.2020.560084. eCollection 2020. PMID 33101174